CLINICAL TRIAL: NCT07336654
Title: Evaluation of a Novel Wearable Device for Circadian Rhythm Monitoring in Healthy, OSA, and Insomnia Participants
Brief Title: Circadian Rhythm Monitoring Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MA250925
Record Dates: First submitted 2026-01-01; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Circadian rhythm monitoring (Experimental): All participants will be provided a wearable non-invasive device which aims to measure circadian rhythm information
  Interventions: Device: Circadian monitoring device

INTERVENTIONS:
Device: Circadian monitoring device — This is a new wearable device for non-invasive continuous monitoring of physiological signals to derive circadian rhythm

SUMMARY:
This will be a single-center, prospective observational study designed to evaluate the feasibility and accuracy of a new wearable device for non-invasive continuous monitoring of physiological signals to derive circadian rhythm. Melatonin sampling will be included for comparison against wearable-derived measures

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years at screening.
* Able and willing to provide written informed consent.
* Belonging to one of three strata: (a) healthy controls without diagnosed sleep disorder, (b) patients with physician-diagnosed OSA, or (c) patients with physician-diagnosed insomnia (based on DSM-5/AASM criteria and ISI ≥15)
* Capable of using a smartphone for app-based data syncing.
* Willing to comply with study visits, wearable use, and saliva sampling.

Exclusion Criteria:

* • Dermatologic conditions preventing wearable use.

  * Significant psychiatric or neurologic illness that may impair compliance.
  * Shift work or trans-meridian travel within 2 weeks prior.
  * Currently pregnant
  * Use of medications known to significantly alter circadian rhythm (e.g., exogenous melatonin, beta-blockers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Association between circadian phase estimated by the wearable device and circadian phase determined by salivary melatonin sampling. | 48 hours
  Data taken from melatonin sampling will be compared with data taken from the wearable device to determine the wearables' ability to estimate circadian phase

IPD SHARING:
Plan to Share IPD: No
Pilot study to determine feasibility only